CLINICAL TRIAL: NCT02337231
Title: Role of Fatty Acid Desaturase(s) (FADS) Polymorphisms in Determining the In Vivo Metabolism of Polyunsaturated Fatty Acids (PUFAs) in Botanical Oils in Humans.
Brief Title: Botanical Oils Study to Determine Genetic Differences in the Way Your Body Processes Fats in Edible Oils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00025085; P50AT002782-08 (NIH)
Record Dates: First submitted 2014-12-17; First posted 2015-01-13 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Genetic Differences of Lipid Metabolism/Healthy Subjects
MeSH Terms: interventions — Soybean Oil; borage oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GG genotype (Other): Healthy participants with genotype GG at rs174537 will take gel capsules that contain soybean oil (4-weeks) and borage oil (4-weeks) in a crossover study.
  Interventions: Dietary Supplement: soybean oil and borage oil
- GT genotype (Other): Healthy participants with genotype GT at rs174537 will take gel capsules that contain soybean oil (4-weeks) and borage oil (4-weeks) in a crossover study.
  Interventions: Dietary Supplement: soybean oil and borage oil
- TT genotype (Other): Healthy participants with genotype TT at rs174537 will take gel capsules that contain soybean oil (4-weeks) and borage oil (4-weeks) in a crossover study.
  Interventions: Dietary Supplement: soybean oil and borage oil

INTERVENTIONS:
Dietary Supplement: soybean oil and borage oil — Compare the capacity of humans with GG, GT and TT genotypes at rs174537 taking soybean and borage oils to metabolize medium chain PUFAs.
  Other Names: Botanical oil

SUMMARY:
A randomized, controlled, cross-over clinical trial of borage oil vs soybean oil to determine whether the metabolism and/or impact of medium chain-polyunsaturated fatty acids (MC-PUFAs) in botanical oil supplements are changed in relationship to specific genotypes in a SNP (rs174537) strongly associated with FADS1 activity and PUFA metabolism.

DETAILED DESCRIPTION:
The study will be a randomized, controlled, cross-over clinical trial of borage oil and soybean oil to determine whether the metabolism and/or impact of MC-PUFAs in botanical oil supplements are changed in relationship to specific genotypes in a SNP (rs174537) strongly associated with FADS1 activity and PUFA metabolism. Subjects previously genotyped at rs174537 will be given supplements and both blood PUFA (serum and erythrocyte membranes), urinary eicosanoids and eicosanoid release from whole blood (leukocyte generation) will be measured as biochemical determinants of genotype impact on supplement metabolism.

To evaluate the effect of genotype at the rs174537 locus on the metabolism of MC-PUFAs in borage and soybean oil to long chain polyunsaturated fatty acids (LC-PUFAs), including arachidonic acid, the investigators will utilize a double blind, randomized, crossover design. There will be three study groups based on the genotype of the healthy volunteer at rs174537. Individuals within each genotype will be consented and screened up to 8 weeks prior to randomization and the start of the intervention. Subjects will be randomized to begin with 4 weeks of either borage oil or soybean oil followed by an 8 week washout period, and then another 4 week period in which they take the second oil. Study visits will occur at 0, 2, and 4 weeks during each oil supplementation period, in addition to the consenting visit, for a total of 7 visits during the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Must agree to adhere to dietary requirements during the entire study
* Be willing to participate for the whole study
* Be willing to not take PUFA supplements outside of those provided by the study
* Agree not to take interfering medications during the duration of the study
* Agree to allow samples to be stored for future use

Exclusion Criteria:

* May not have diabetes, cancer, heart attack or vascular surgery within the past year, be diagnosed with heart disease, have uncontrolled high blood pressure, history of stroke, atherosclerosis, asthma, multiple sclerosis or chronic joint disease
* Gallbladder removal or gallbladder disease
* Use of tobacco products within the last six months
* Pregnancy or lactation
* Fasting triglycerides greater than 150 mg/dl
* Blood pressure greater than 130/90
* BMI equal to or greater than 30 or less than 19
* Fasting glucose greater than 125 mg/dl
* Have liver function values in the normal range
* Taking greater than 100 mg aspirin/day
* Taking NSAIDS or oral corticosteroids
* Taking montelukast-type allergy medications
* Having a pacemaker or a defibrillator
* Taking lipid lowering medications

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Change in serum fatty acids from baseline as measured in mass and recorded as mg/dL | 16-week study

CONTACTS AND LOCATIONS:
Overall Officials: Floyd H. Chilton, Ph.D., Principal Investigator — Wake Forest Health Science; Priscilla Ivester, M.S., Study Chair — Wake Forest Health Science; Tammy Lee, M.S., Study Chair — Wake Forest Health Science; Susan Sergeant, Ph.D., Study Director — Wake Forest Health Science
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Study recruitment has just been completed. Samples are beginning to be analysed and data will be shared when available

REFERENCES:
- [Derived] Sergeant S, Hallmark B, Mathias RA, Mustin TL, Ivester P, Bohannon ML, Ruczinski I, Johnstone L, Seeds MC, Chilton FH. Prospective clinical trial examining the impact of genetic variation in FADS1 on the metabolism of linoleic acid- and ɣ-linolenic acid-containing botanical oils. Am J Clin Nutr. 2020 May 1;111(5):1068-1078. doi: 10.1093/ajcn/nqaa023. PMID 32167131